CLINICAL TRIAL: NCT03072225
Title: Randomized Controlled Clinical Study on Vulnerable Plaque of Carotid Artery With Chinese Herbal and Insects Medicine
Brief Title: Study on Vulnerable Plaque of Carotid Artery With Chinese Herbal and Insects Medicine
Acronym: Spchim
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YN2014LN08
Record Dates: First submitted 2017-02-18; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Carotid Artery Plaque
Keywords: herbal medicine; stroke; vulnerable plaques of carotid artery
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal Medicine C-117 (Experimental): Herbal Medicine C-117 Prescription (6g/bag，one bag each time, twice a day.) for 6 months
  Interventions: Drug: Herbal Medicine C-117
- The Placebo of Herbal Medicine C-117 (Placebo Comparator): Placebo of Herbal Medicine C-117 (6g/bag，one bag each time, twice a day.) for 6 months
  Interventions: Drug: The Placebo of Herbal Medicine C-117

INTERVENTIONS:
Drug: Herbal Medicine C-117 — Herbal Medicine C-117 formula including 2 herbals and 2 insects
  Arms: Herbal Medicine C-117
Drug: The Placebo of Herbal Medicine C-117 — The Placebo of Herbal Medicine C-117 formula including 4 herbals
  Arms: The Placebo of Herbal Medicine C-117

SUMMARY:
The investigators want treat Vulnerable plaque of carotid artery with a herbal and insects Chinese medicine. Designing a RCT trial to prove the effect and safety.

DETAILED DESCRIPTION:
Vulnerable plaque of carotid artery is the important intervention target for primary prevention and secondary prevention of cerebral arterial thrombosis, but there are no effective, safe and prevalent treatment measures against it. The development that traditional Chinese medicine has achieved in treating plaque of carotid artery shows that great accomplishment could be made within this area. Academia should engage in clinical research on regulated treatment methods in traditional Chinese medicine with long-term intervention and high patient compliance, providing strong evidence for evidence-based medicine and guidance to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of carotid artery atherosclerosis;
2. Ultrasound of carotid artery atherosclerosis plaque specifies it as unstable plaque (including malacoplakia and mixed plaque);

Exclusion Criteria:

1. mRS Rating higher than or equal to 3 before joining the trail group;
2. Carotid artery stenosis is higher than or equal to 50%;
3. Confirmed as or suspected to be vasculitis;
4. With infection, tumor or insufficient heart, liver and kidney functions (renal function higher than twice of upper limit in normal limit, HYHA heart function grading higher than or equal to level 2 );
5. With acute myocardial infarction and unstable angina pectoris;
6. With acute cerebral arterial thrombosis;
7. lesion: Severe stenosis or occlusion of distal intracranial vessels;
8. Pregnant women or lactating mothers;
9. With known history of allergy to the drugs of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The total number of all-cause mortality and all-cause stroke within 12 months | 1 years
  After drug-use 6 months, observe all-cause mortality and all-cause stroke (hemorrhage or ischemic).

SECONDARY OUTCOMES:
The nature of Vulnerable plaque of carotid artery through color ultrasound | 6 months
  At the time of 6 months, observe the nature of Vulnerable plaque of carotid artery through color ultrasound, comparing with the result before using drugs
The number of Vulnerable plaque of carotid artery through color ultrasound | 6 months
  At the time of 6 months, observe the nature of Vulnerable plaque of carotid artery through color ultrasound, comparing with the result before using
Blood lipid levels | 6 months
  At the time of 6 months, the investigators will observe the blood lipid levels

CONTACTS AND LOCATIONS:
Overall Officials: Jianwen Guo, MD, Principal Investigator — Guangdong Province Hospital of Tradtional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong B, Chen X, Lin R, Zhang F, Zhong J, Zhang Q, Zhou Y, Li H, Zeng L, Jiang Z, Guo J. Safety and Efficacy of the C-117 Formula for Vulnerable Carotid Artery Plaques (Spchim): A Randomized Double-Blind Controlled Pilot Study. Evid Based Complement Alternat Med. 2019 Jul 17;2019:9746492. doi: 10.1155/2019/9746492. eCollection 2019. PMID 31391862